CLINICAL TRIAL: NCT03353337
Title: A Randomised Controlled Trial of Aerobic Exercise for Inpatients With Bipolar Affective Disorder
Brief Title: A Study of Aerobic Exercise for Patients With Bipolar Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Psychiatric Hospital (Other Government)
Responsible Party: Principal Investigator, Kangguang Lin, MD,PhD, Guangzhou Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GZ Psychiatric Hospital
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Bipolar Disorder; Cognitive Symptom
Keywords: neurocognition; prognosis; aerobic exercise
MeSH Terms: conditions — Bipolar Disorder; Neurobehavioral Manifestations | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic exercise (Experimental): Cycling at the intensity of 50%-70% of maximum heart rate (220-age) for 30 mins per day, 4 days per week, last for 1 month.
  Interventions: Behavioral: aerobic exercise
- Placebo controlled group (Placebo Comparator): General intensity activities of recreation therapy, including Handicraft manufacture, reading activity, singing entertainment, walking.
  Interventions: Behavioral: Placebo controlled group

INTERVENTIONS:
Behavioral: aerobic exercise — Cycling at the intensity of 50%-70% of maximum heart rate (220-age) for 30 mins per day, 4 days per week, last for 1 months.
  Arms: aerobic exercise
Behavioral: Placebo controlled group — General intensity activities of recreation therapy, including Handicraft manufacture, reading activity, singing entertainment, walking.
  Arms: Placebo controlled group

SUMMARY:
This study will investigate the effects of aerobic exercise on mental states, cognition, BDNF, and long-term outcomes in patients with bipolar disorder.

DETAILED DESCRIPTION:
Multiple cognitive impairments are common in patients with bipolar disorder. Preliminary evidence shows that aerobic exercise might have positive effects in enhancing cognition and improving clinical symptoms in patients with mood disorders. This randomized controlled trial will investigate short-term (1 months) effects of aerobic exercise on cognition and clinical symptoms as well as the long-term (12 months) effects on decreasing the recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV defined bipolar disorder.
* Never accept aerobic exercise therapy.
* dextromanuality.

Exclusion Criteria:

* Diagnosed neurological or musculoskeletal disorder/injury,
* Uncontrolled cardiovascular or metabolic diseases that are not suitable for running
* Diagnosed hypertension
* Other diagnosed serious medical conditions that are not suitable for cycling
* Severe suicidal ideation
* Mental retardation
* Currently participating in a exercise program or activity, defined as 30 minutes of vigorous physical activity 4-5 times per week

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in neurocognitive function | 12 months
  Changes in neurocognitive function measured by the MATRICS Consensus Cognitive Battery (MCCB) after three months (12 weeks) of aerobic exercise
Changes in neurocognitive function | Changes in neurocognitive function measured by the MATRICS Consensus Cognitive Battery (MCCB) after three months (12 weeks) of aerobic exercise
  Changes in neurocognitive function measured by the MATRICS Consensus Cognitive Battery (MCCB) after three months (12 weeks) of aerobic exercise

SECONDARY OUTCOMES:
relapse rate | 12 months
  Relapses of depressive and/or hypo/manic episodes
depressive symptoms | 4 weeks, 4 months, 12 months
  depressive symptoms measured by Hamilton Depression Scale
manic symptom | 4 weeks, 4 months, 12 months
  manic symptom measured by Young Manic Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Kangguang Lin, MD, PhD, Principal Investigator — Guangzhou Brain hospital (Guangzhou Psychiatric Hospital)
Locations (1):
- Guangzhou Brain hospital(Guangzhou Huiai Hospital), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided